Study flow chart

ClinicalTrials.gov NCT03176056

Unique Protocol ID: 201504032RINA

Brief Title: The Effectiveness of Low Carbohydrate Diet in Reducing Polypharmacy for

Patients With Type 2 Diabetes Mellitus

Official Title: Low Carbohydrate Diet for Type 2 Diabetes Mellitus

July, 31. 2016

